CLINICAL TRIAL: NCT00078442
Title: A Phase II Open-Label Pilot Trial of the Antiretroviral Activity, Safety, and Tolerability of Pegylated Interferon Alfa-2A (40KD) [PegasysTM] in HIV-1 Infected Subjects
Brief Title: Safety and Tolerability of Pegylated Interferon (PEG-IFN) Alfa-2a in HIV Infected People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5192; DAIDS-ES ID 10013
Record Dates: First submitted 2004-02-25; First posted 2004-02-26 (Estimated); Last update posted 2009-08-07 (Estimated); Status verified 2009-08

CONDITIONS: HIV Infections
Keywords: Treatment Experienced; Treatment Interruption; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — peginterferon alfa-2a

ARMS (1):
- 1 (Experimental): Participants will receive weekly injections of 180 mcg PEG-IFN alfa-2a at the clinic for 12 weeks. After Week 12, participants will be followed off-treatment until Week 18.
  Interventions: Drug: Pegylated interferon alfa-2a

INTERVENTIONS:
Drug: Pegylated interferon alfa-2a — Recombinant PEG-IFN alfa-2a is a synthetic version of IFN and is used in hepatitis C virus treatment

SUMMARY:
Recombinant interferon (IFN) may be useful in the treatment of HIV. However, the high doses of IFN necessary to keep HIV under control limit its use due to toxic side effects. The purpose of this study is to test the safety and tolerability of weekly recombinant pegylated interferon (PEG-IFN) alfa-2a in HIV infected people who are currently on antiretroviral therapy (ART) interruption or who have not started taking anti-HIV drugs.

DETAILED DESCRIPTION:
IFN is an immune response enhancer and is produced in the body in response to viral infection. PEG-IFN may have less harmful side effects than non-pegylated IFN. Recombinant PEG-IFN alfa-2a is a synthetic version of IFN and is used in hepatitis C virus treatment. PEG-IFN alfa-2a has demonstrated potentially useful antiviral properties in HIV treatment; however, due to the high doses that must be administered to maintain viral suppression, toxicity (especially to the blood) is a concern. This study will evaluate the safety, tolerability, and antiretroviral activity of PEG-IFN alfa-2a in HIV infected patients who have received ART in the past but are currently off ART or who are ART naive.

The study will last 18 weeks. Participants will receive weekly injections of 180 mcg PEG-IFN alfa-2a at the clinic for 12 weeks. After Week 12, participants will be followed off-treatment until Week 18. Physical exams will be performed weekly. Blood collection to monitor viral load, PEG-IFN alfa-2a serum levels, and CD4 and CD8 counts will be conducted at selected weeks during the study. Filgrastim will be given to patients who exhibit neutropenic toxicity.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count of 300 cells/ml or greater within 30 days of study entry
* HIV viral load of 5000 copies/ml or greater within 30 days of study entry
* Received ART previously but have currently interrupted treatment within 12 weeks prior to study entry OR ART naive
* Willing to delay initiation or re-initiation of antiretroviral medications for the duration of the study
* Agree to use acceptable forms of contraception

Exclusion Criteria:

* Previous use of interferon alfa
* Known allergy or sensitivity to PEG-IFN alfa-2a or its formulation
* Active drug or alcohol abuse that would interfere with the study
* Acute therapy for a serious infection within 30 days of study entry
* Use of non-protocol-specified immunomodulatory therapy within 60 days of study entry
* Active immunization within 30 days of study entry
* History of severe psychiatric disease such as major depression, suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to psychiatric disease
* History of poorly controlled thyroid disease, including history of elevated thyroid stimulating hormone (TSH) levels with elevated antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease
* History of clinically significant heart disease that could be worsened by acute anemia
* History of severe seizure disorder or current anticonvulsant use
* Hepatitis C antibody positive within 60 days prior to study entry
* Hepatitis B surface antigen positive within 60 days prior to study entry
* Known sensitivity to E. coli derived products, such as filgrastim
* Any past evidence of chronic liver disease
* Any past or current evidence of immunologically-mediated disease
* Evidence of chronic pulmonary disease
* Severe eye problems due to diabetes, hypertension, cytomegalovirus infection, or macular degeneration
* History of major organ transplantation with an existing functional graft
* History or other evidence of severe illness, cancer, or other conditions that would make the patient unsuitable for the study
* Hemoglobin abnormalities or any other cause of or tendency for breakdown of red blood cells
* Any medical condition that would prevent successful completion of the study
* Use of certain medications
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-05; Primary Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
CD4 count | Throughout study
CD8 count | Throughout study
Laboratory and clinical adverse effects | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: David Asmuth, MD, Study Chair — Division of Infectious and Immunologic Diseases, University of California, Davis Medical Center
Locations (3):
- United States (3):
  - University of California, Davis Medical Center, Sacramento, California
  - Northwestern University, Chicago, Illinois
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Bain VG. Effect of HCV viral dynamics on treatment design: lessons learned from HIV. Am J Gastroenterol. 2001 Oct;96(10):2818-28. doi: 10.1111/j.1572-0241.2001.04234.x. PMID 11693314
- [Background] Dwyer JT, Paul SM. HIV and hepatitis C co-infection. N J Med. 2003 Sep;100(9 Suppl):50-4; quiz 77-8. PMID 14556604
- [Background] Emilie D, Burgard M, Lascoux-Combe C, Laughlin M, Krzysiek R, Pignon C, Rudent A, Molina JM, Livrozet JM, Souala F, Chene G, Grangeot-Keros L, Galanaud P, Sereni D, Rouzioux C; Primoferon A Study Group. Early control of HIV replication in primary HIV-1 infection treated with antiretroviral drugs and pegylated IFN alpha: results from the Primoferon A (ANRS 086) Study. AIDS. 2001 Jul 27;15(11):1435-7. doi: 10.1097/00002030-200107270-00014. PMID 11504966
- [Background] Kawakami K. Promising immunotherapies with Th1-related cytokines against infectious diseases. J Infect Chemother. 2003 Sep;9(3):201-9. doi: 10.1007/s10156-003-0263-5. PMID 14513386
- [Background] Levy JA, Scott I, Mackewicz C. Protection from HIV/AIDS: the importance of innate immunity. Clin Immunol. 2003 Sep;108(3):167-74. doi: 10.1016/s1521-6616(03)00178-5. No abstract available. PMID 14499239
- [Derived] Asmuth DM, Murphy RL, Rosenkranz SL, Lertora JJ, Kottilil S, Cramer Y, Chan ES, Schooley RT, Rinaldo CR, Thielman N, Li XD, Wahl SM, Shore J, Janik J, Lempicki RA, Simpson Y, Pollard RB; AIDS Clinical Trials Group A5192 Team. Safety, tolerability, and mechanisms of antiretroviral activity of pegylated interferon Alfa-2a in HIV-1-monoinfected participants: a phase II clinical trial. J Infect Dis. 2010 Jun 1;201(11):1686-96. doi: 10.1086/652420. PMID 20420510